CLINICAL TRIAL: NCT01588223
Title: A Non Invasive Diagnostic of Endometrial Receptivity Based on Lipidomic Profile on Endometrial Fluid.
Brief Title: Non Invasive Diagnostic of Endometrial Receptivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Igenomix (Industry)
Responsible Party: Principal Investigator, Carlos Simon, Prof. Carlos Simon, MD PhD, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1002-C-069-OB
Record Dates: First submitted 2012-04-26; First posted 2012-04-30 (Estimated); Last update posted 2014-03-27 (Estimated); Status verified 2014-03

CONDITIONS: Endometrial Receptivity Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lipids (Experimental)
  Interventions: Other: Lipid identification

INTERVENTIONS:
Other: Lipid identification — The lipids are identified using Mass Spectrometry

SUMMARY:
The purpose of this study is to determine a lipidomic profile on the endometrial fluid, that can predict endometrial receptivity.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors undergoing controlled ovarian stimulation
* Regular menstrual cycles
* no abnormal karyotype
* generally healthy
* BMI 19-29 Kg/m2 (both inclusive)
* 18 to 35 years old.

Exclusion criteria:

-patients diagnosed with endometriosis and/or endometritis.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Levels of lipids in the endometrial fluid as a diagnostic factor. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Spain